CLINICAL TRIAL: NCT01735331
Title: Vascular Endothelial Growth Factor Levels at Hysteroscopic Biopsies Which Taken From Recurrent Pregnancy Loss
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: BEHGynObs-3
Record Dates: First submitted 2012-11-26; First posted 2012-11-28 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Recurrent Pregnancy Loss Without Current Pregnancy
Keywords: Vascular endothelial growth factor, Recurrent Pregnancy Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VEGF level: VEGF level in hysteroscopic endometrial biopsy of the patients with recurrent pregnancy loss.
- control group: Patients with Abnormal Uterine Bleeding

SUMMARY:
The aim of this study is determine vascular endothelial growth factor levels and angiogenesis/vascularity from hysteroscopic endometrial biopsies which taken from patients who has Recurrent Pregnancy Loss.The endometrial vascular endothelial growth factor levels will be measured by immunohistochemical staining methods due to office hysteroscopic endometrial biopsy after the menstruation at follicular phase of menstrual cycle.

DETAILED DESCRIPTION:
This study is a prospective,observational,single-center study.Ethical approval was obtained from the Institutional Review Board.This study will be completed 30 patients with Habitual Abortus.

Endometrial vascular endothelial growth factor levels will be measured using Flk-1 / Kinase Domain Receptor / Vascular endothelial growth factor receptor-2, Ab-1 (Rabbit PAb), Vascular Endothelial Growth Factor (VEGF) Ab-7 (VG1), Cluster of Differentiation 34 (Endothelial Cell Marker) Ab-1 (QBEnd/10), Vascular endothelial growth factor receptor-1 (N-term) (FLT1) antibody kits. All assays will be performed according to the manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Recurrent Pregnancy Loss who accept to join the study.

Exclusion Criteria:

* Patients whose age of <18 and >45
* Patients with have any pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patients with Recurrent Pregnancy Loss
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of this study is to determine endometrial vascular endothelial growth factor levels in patient with Recurrent Pregnancy Loss | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: TANER A. USTA, M.D., Principal Investigator — Bagcilar Training and Research Hospital,Istanbul,Turkey.
Locations (1):
- Bagcilar Training and Research Hospital, Istanbul, Turkey (Türkiye)